CLINICAL TRIAL: NCT03273803
Title: Cardiac Auscultation Using Smartphones: a Proof-of-concept Study
Brief Title: Cardiac Auscultation Using Smartphones
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Advanced Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Jung-Won Suh, MD, PhD, Seoul National University Hospital
Other Study IDs: B-1609-361-303
Record Dates: First submitted 2017-09-03; First posted 2017-09-06 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Cardiovascular Physiological Phenomena
Keywords: Heart sounds, smartphone, application

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Heart sound recording using smartphone application — Heart sound recording and analysis using android smartphones (Samsung Galaxy S5, Galaxy S6, and LG G3)

SUMMARY:
The investigators performed a proof-of-concept study enrolling subjects with normal and pathologic heart sounds. Heart sound was recorded by auscultation on the skin of the chest wall using three smartphones: Samsung Galaxy S5 and Galaxy S6, and LG G3 . Recorded heart sounds were processed and classified by a diagnostic algorithm using convolutional neural networks.

DETAILED DESCRIPTION:
Heart sound recording was done by researchers who were familiar with the use of the app and understand the principles of cardiac auscultation.

Reference heart sounds were recorded using an electronic stethoscope (3M™ Littmann® Electronic Stethoscope Model 3200). Study devices included Samsung Galaxy S5 (model SM-G900), Galaxy S6 (SM-G920), and LG G3 (LG-F400).

ELIGIBILITY:
Inclusion Criteria:

* subjects who gave informed consent
* subjects who are 18 years old or older and had performed ECG and echocardiography during the previous 6 months.

Exclusion Criteria:

* subjects with impairment of cognition

Age Groups: Child, Adult, Older Adult
Study Population: Men and women were evenly enrolled, and the median age was 65.5 years.
  Twenty subjects (43.5%) had systolic murmur, 20 (43.5%) normal heart sound, 5 (10.9%) diastolic murmur, and 1 (2.2%) S4.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of "CPstethoscope" in interpretation of heart sounds | 0
  specificity, sensitivity, negative predictive value, positive predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Won Suh, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang SH, Joe B, Yoon Y, Cho GY, Shin I, Suh JW. Cardiac Auscultation Using Smartphones: Pilot Study. JMIR Mhealth Uhealth. 2018 Feb 28;6(2):e49. doi: 10.2196/mhealth.8946. PMID 29490899